CLINICAL TRIAL: NCT02356146
Title: First Tacrolimus Dose Trough Level is Better Than CYP3A5 Genotyping in Tacrolimus Dose Prediction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Natavudh Townamchai, MD, Assistant Professor, Chulalongkorn University
Other Study IDs: IRB225/56
Record Dates: First submitted 2015-02-01; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Kidney Transplantation Recipients
Keywords: Kidney transplantation; genotype; tacrolimus; CYP3A5

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood level for tacrolimus was took 12 hours after first dose.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All KT recipient
  Interventions: Drug: Tacrolimus C12

INTERVENTIONS:
Drug: Tacrolimus C12

SUMMARY:
Tacrolimus dose highly varies among Asian kidney transplant recipients. This can be explained by variety of CYP3A5 expression. CYP3A5 genotyping is highly recommended for patients receiving tacrolimus. Here, we assessed the tacrolimus dose prediction by comparing CYP3A5 expression and tacrolimus dosage using tacrolimus concentration after single dose administration prior to kidney transplantation.

Plasma tacrolimus trough level was measured at 12 hours after first dose of 0.1 mg/kg of tacrolimus (TacC12), orally administered in 51 new kidney transplant recipients. Patients with CYP3A5 inhibitor/inducer co-medications were excluded. Genotyping for CYP3A5 expression were carried out by RT-PCR. The dosages of tacrolimus at post-operative day 7 and dosage which provided stable therapeutic levels in post-operative month 1 to 3 (C0 5-8 ng/mL) were recorded.

The genotyping, TacC12, and target tacrolimus dosage have good correlations.

ELIGIBILITY:
Inclusion Criteria:

* All KT recipients

Exclusion Criteria:

* Recipient who not receiving tacrolimus

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All KT recipient who transplanted and will be transplanted in King Chulalongkorn Memorial Hospital from 2012-2015
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
target tacrolimus dose at 3 months | 3 months

SECONDARY OUTCOMES:
rate of rejection | 3-12 months
rate of CNI toxicity | 2-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Natavudh Townamchai, MD, Principal Investigator — Chulalongkorn University and King Chulalongkorn Memorial Hospital, Thai Red Cross Society
Locations (1):
- Chulalongkorn University and King Chulalongkorn Memorial Hospital, Bangkok, Thailand